CLINICAL TRIAL: NCT04804566
Title: Understanding Fabry Disease Therapy Choices Through the Eyes of the Patients
Status: Completed | Type: Observational
Sponsor: Amicus Therapeutics (Industry)
Collaborators: Engage Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AT-NIS-00002
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Fabry Disease
Keywords: Hypohidrosis; Proteinuria; Angiokeratoma
MeSH Terms: conditions — Fabry Disease; Hypohidrosis; Proteinuria; Angiokeratoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- ERT User- Did Not Switch to Galafold: ERT users with mutation amenable to Galafold who did not switch
  Interventions: Other: This is a non-interventional study
- ERT User- Switched and Stayed on Galafold: ERT users with the mutation amenable to Galafold who switched and stayed on Galafold
  Interventions: Other: This is a non-interventional study
- No Previous Therapy- Started Galafold and Stayed On: Those naïve to therapy with the mutation amenable to Galafold who went on and stayed on Galafold
  Interventions: Other: This is a non-interventional study
- No Previous Therapy- No Current Therapy: Those who were naïve to therapy with the mutation amenable to Galafold and have never been on any therapy.
  Interventions: Other: This is a non-interventional study
- ERT Users- Switched and Discontinued Galafold: Participants who are ERT users with an amenable mutation who switched to and later discontinued Galafold
  Interventions: Other: This is a non-interventional study
- No Previous Therapy- Started Galafold and Discontinued: Participants who are naïve to therapy with an amenable mutation, went on Galafold, and discontinued
  Interventions: Other: This is a non-interventional study

INTERVENTIONS:
Other: This is a non-interventional study — This is a non-interventional study

SUMMARY:
The objective of this study is to increase the understanding surrounding the choices presented to patients and families impacted by Fabry disease.

DETAILED DESCRIPTION:
This will be a cross-sectional study conducted in approximately 130 individuals (or representative parents/caregivers of patients) living with Fabry disease. All study participants will complete the RSVP followed by a structured interview conducted by trained interviewers. It is estimated that each respondent will need up to 60 minutes for the entire process; 10 minutes to complete the RSVP including uploading the proof of Fabry disease diagnosis or verifying membership with Fabry groups, including but not limited to: Fabry Support and Information Group, National Fabry Disease Foundation, MPS Society UK, Morbus Fabry Selbsthilfergruppe, Fabry International Network, or others, and approximately 50 minutes to complete the interview.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a person with Fabry disease who is 18 years or older or the parent/legal guardian of a living person with Fabry disease who is under the age of 18 years or who are 18 years and older who are unable to answer for themselves.
* Confirmed diagnosis of Fabry disease with written proof of disease provided
* Must have a genetic mutation that is amenable to oral therapy
* Resident of Germany, the U.K or the U.S.
* Able to read, write and communicate in German, or English.
* Able to grant informed consent
* Willing to participate in a 50 to 60-minute telephone interview, including follow up questions (if necessary) and information regarding adverse events (if necessary).

Exclusion Criteria:

* Inability to meet any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Purposive sampling techniques will be used which will seek to initially recruit 30 participants (person with Fabry or their parent/legal guardian) from each of four groups noted below:
  1. ERT users with an amenable mutation, who did not switch
  2. ERT users with an amenable mutation, who switched to Galafold and stayed on
  3. Those naïve to therapy with an amenable mutation, who went on Galafold and stayed on
  4. Those naïve to therapy with an amenable mutation, who have never been on any therapy.
  There will also be an attempt to recruit 5 patients from each of the two groups:
  1. ERT users with an amenable mutation, who switched and discontinued Galafold, and
  2. Those naïve to therapy, with an amenable mutation, who went on Galafold and discontinued.
  In order to get a geographic sampling, the first four groups will attempt to recruit 30 patients/parents or caregivers of patients with representation from Germany, the UK, and the US.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Patterns and Trends that Provide Evidence and Context for the Treatment Choices and Experiences of Those with Fabry Disease | 1-2 months
  The goal of the statistical analysis is to uncover patterns and trends that provide both evidence and context for the treatment choices and experiences of patients and families impacted by Fabry disease.
  All findings will be summarized in the final report, which will not identify any respondent as described above. At the conclusion of this study, the researchers may publish their findings in a medical / scientific journal.

CONTACTS AND LOCATIONS:
Overall Officials: Niloofar Nobakht, MD, Principal Investigator — Ronald Regan UCLA Medical Center
Locations (1):
- Engage Health, Eagan, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The pseudonymized answers provided by each respondent will be combined with those of others participating in the study and the pseudonymized database (Excel format) will be locked and provided to Engage Health personnel for analysis ("Study Data"). The goal of the statistical analysis is to uncover patterns and trends that provide both evidence and context for the treatment choices and experiences of patients and families impacted by Fabry disease.
  All findings will be summarized in the final report, which will not identify any respondent as described above. At the conclusion of this study, the researchers may publish their findings in a medical/scientific journal.
Supporting Information: SAP, Analytic Code

REFERENCES:
- See also: Galafold and Fabry Disease — https://www.galafold.com/fabry-disease.php
- See also: Review of Fabry Disease — https://www.ncbi.nlm.nih.gov/pubmed/29562089